CLINICAL TRIAL: NCT05688969
Title: Mechanisms of Anabolic Osteoporosis Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1P50AR080596-01 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: 1:1 allocation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Biopsy (Active Comparator): The investigators will perform paired iliac crest bone biopsies in postmenopausal women who meet standard romosozumab treatment indications and are being prescribed romosozumab by their treating physician. All study volunteers will have a bone biopsy procedure prior to starting therapy, and then an identical procedure at the contralateral side either 3-6 weeks ("early") or 6-8 months ("late") after starting therapy. This is not a clinical trial: the investigators will not be assigning volunteers to a specific osteoporosis therapy, though the investigators will randomize volunteers to either the early or late second biopsy.
  Interventions: Other: early versus late biopsy
- Late Biopsy (Active Comparator): The investigators will perform paired iliac crest bone biopsies in postmenopausal women who meet standard romosozumab treatment indications and are being prescribed romosozumab by their treating physician. All study volunteers will have a bone biopsy procedure prior to starting therapy, and then an identical procedure at the contralateral side either 3-6 weeks ("early") or 6-8 months ("late") after starting therapy. This is not a clinical trial: the investigators will not be assigning volunteers to a specific osteoporosis therapy, though the investigators will randomize volunteers to either the early or late second biopsy.
  Interventions: Other: early versus late biopsy

INTERVENTIONS:
Other: early versus late biopsy — early (3-6 weeks) versus late (6-8 months) biopsy

SUMMARY:
The aim of this study is to investigate the effect of romosozumab on bone cells during early and late phases of treatment.

DETAILED DESCRIPTION:
The investigators will perform paired iliac crest bone biopsies in postmenopausal women who meet standard romosozumab treatment indications and are being prescribed romosozumab by their treating physician. All study volunteers will have a bone biopsy procedure prior to starting therapy, and then an identical procedure at the contralateral side either 3-6 weeks ("early") or 6-8 months ("late") after starting therapy. This is not a randomized clinical trial testing the efficacy of a drug - the investigators will not be assigning volunteers to a specific osteoporosis therapy, though the investigators will randomize volunteers to either the early or late second biopsy.

ELIGIBILITY:
Inclusion Criteria:

All postmenopausal women who are prescribed romosozumab by their treating physicians, meet the FDA-defined indication for romosozumab, and who are not at increased risk for a bone marrow aspirate or bone biopsy will be offered enrollment. The FDA approved indication for romosozumab is: "the treatment of osteoporosis in postmenopausal women at high risk for fracture, defined as a history of osteoporotic fracture, or multiple risk factors for fracture; or patients who have failed or are intolerant to other available osteoporosis therapy." Volunteers must be:

1. Female aged > 45 years
2. Postmenopausal by either of the following criteria:

   1. > 36 since last spontaneous menses
   2. > 36 months since hysterectomy, plus serum FSH > 40 units / liter if < 60 years

Exclusion Criteria:

* renal disease (stage 4 CKD)
* elevated blood PTH (intact PTH > 77 pg/ml).
* serum 25-OH vitamin D < 20 ng/ml
* major psychiatric disease that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
* excessive alcohol use or substance abuse that would preclude the subject from providing adequate informed consent or completing the protocol procedures.
* known congenital or acquired bone disease other than osteoporosis.
* exposure to oral bisphosphonates within the past 3 months, denosumab in the last 12 months, intravenous bisphosphonates within the past 24 months.
* exposure to estrogens, SERMs, or calcitonin, oral or parenteral glucocorticoids for more than 14 days in the past 2 months.
* any prior exposure to romosozumab.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 16 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Osteoblast progenitor cell numbers | 3-6 weeks (early) versus 6-8 months (late)
  The investigators are testing the mechanistic hypothesis that romosozumab treatment increases osteoblast progenitor cell numbers at early, but not late, treatment time points.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States